CLINICAL TRIAL: NCT00109018
Title: Nitrite as a Marker of Cardiovascular Risk; Development of Novel Biomarkers in Patients With Coronary Artery Disease
Brief Title: Biomarkers for Cardiovascular Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050145; 05-H-0145
Record Dates: First submitted 2005-04-21; First posted 2005-04-22 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-04-15

CONDITIONS: Coronary Artery Disease
Keywords: Risk Assessment; Coronary Heart Disease; Vascular Function; Nitric Oxide Metabolites; Blood Tests; Nitrite; Flow-Mediated Dilation; Biomarker; Endothelial Dysfunction; Coronary Artery Disease; CAD; Coronary Artery Disease At Risk; Healthy Volunteer
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease

SUMMARY:
Biomarkers for Cardiovascular Disease

Summary: This study will examine the function of the lining cells of blood vessels and measure substances in the blood to see how they relate to various blood tests, including new tests under development to determine cardiovascular disease risk. Nitric oxide is a molecule produced by healthy blood vessels that helps keep them relaxed. Nitrate is a substance formed from nitric oxide in the blood. The release of nitric oxide by blood vessels is reduced in patients with coronary artery disease, compared with healthy people. Also, blood nitrite levels rise in some of these patients. Other substances in the blood and urine also change with risk for heart disease. This study will measure nitrite levels and other inflammatory substances in the blood and urine.

Healthy volunteers, people with various risk factors for heart disease, and people with blockage of one or more major heart arteries or a history of heart attack may be eligible for this study. Candidates must be 21 years of age or older. People who have an irregular heart rhythm or who cannot take oral nitrates are excluded.

Participants undergo the following tests and procedures:

* Blood tests: Samples are drawn three times for routine tests and to look for certain proteins that may affect the heart. Samples are collected once before any other tests, once before starting the exercise stress test (see below) and again after the stress test.
* Urine test: A sample may be tested for proteins in the urine and for other research studies.
* Brachial artery reactivity study: This ultrasound study tests how well a person's arteries widen. The subject rests on a bed. An ultrasound measuring device is placed over the artery just above the elbow. The size of the artery and blood flow through it are measured before and after inflating a pressure cuff around the forearm. The pressure cuff stops the flow of blood to the arm for 5 minutes and then is released while more ultrasound pictures are taken. After the subject rests, a nitroglycerin tablet (medicine that causes blood vessels to relax) is placed under the tongue. After the nitroglycerin is given, the size of the artery and blood flow through it are measured again. After a rest period, the study will be repeated in the healthy volunteers and first 20 patients with heart disease.
* Echocardiography (heart ultrasound): This test involves holding a small probe against the chest to use sound waves for obtaining pictures of the heart. A small catheter (plastic tube) may be placed in a vein to inject a contrast agent that enhances the pictures.
* Metabolic stress testing: Subjects will be asked to breathe in and out of a mask while baseline measurements are taken. Then they exercise on a treadmill while wearing a breathing mask. This test shows how much oxygen the body uses at rest and with exercise.
* Genetic testing (optional): A blood sample is collected to examine DNA - genetic material that determines inherited traits and contains information about body proteins. Some parts of DNA may be used as markers of the level of damage produced by oxygen by-products that may reflect the extent of heart disease in patients. Also, gene variations may make an individual more likely to develop a heart problem. Such markers may guide doctors in predicting how fast the disease will progress or may help find a new type of drug to prevent disease.
* Time requirements: This study is expected to take approximately 5-6 hours for completion within one or two days.
* Follow-up: Patients are contacted by phone every 6 months for information on chest pain, surgical procedures related to the heart, and hospitalizations.

DETAILED DESCRIPTION:
Cardiovascular events are a major cause of morbidity and mortality world-wide and traditional risk factor assessment is limited in its ability to predict which patients will have an event. The endothelium is known to play a central role in vascular homeostasis and nitric oxide (NO) is believed to be the main component responsible for normal endothelial function. Increasing evidence suggests that oxidative stress leading to reduced NO bioavailability and subsequent endothelial dysfunction is an important factor in the progression of vascular diseases. Further investigation of NO metabolites in blood may provide insight into the mechanisms of endothelial dysfunction and disease progression. Preliminary data suggest that although plasma nitrite levels are decreased in CAD patients and correlate with endothelial dysfunction, the nitrite within red blood cells and whole blood is compensatorily increased. Since this new measure is more reproducible and convenient to measure, it may serve as a biomarker of endothelial dysfunction. A prospective study of nitrite and other novel NO-based assays, proteomics, and current biomarkers linked to endothelial function phenotype will allow further investigation into the pathophysiology of endothelial dysfunction and permit development of future markers of atherothrombosis.

ELIGIBILITY:
* INCLUSION CRITERIA

Adults older than 21, of both sexes:

The initial study group will consist of 120 subjects, which will consist of 100 subjects with documented CAD (by cardiac catheterization showing greater than or equal to 70% stenosis in an epicardial vessel), previously documented MI (based on ECG or cardiac enzymes) or CAD risk equivalents (diabetes, peripheral vascular disease, abdominal aortic aneurysm, symptomatic carotid disease, or multiple risk factors that confer a 10 year risk of greater than 20% as defined by the Framingham Risk Score) and 20 healthy age- and sex-matched controls.

Written informed consent.

EXCLUSION CRITERIA

Atrial fibrillation

Any contraindications to oral nitrates

Hypotension, bradycardia.

Myocardial infarction within the prior 30 days

Symptoms of acute CHF

Pregnant women

Receiving active treatment for cancer

Any other condition that may interfere with the interpretation of the study results or not be in the best interest of the subject in the opinion of the investigator.

Since oral nitrate therapy is known to affect serum and possibly whole blood nitrite levels, we will exclude patients on long-acting nitrates for the initial group of 100 cardiac patients. Those patients on chronic nitrate therapy will subsequently be included in the later portion of the study but will be analyzed separately.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2005-04-19; Study Completion 2009-04-15

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Myerburg RJ, Interian A Jr, Mitrani RM, Kessler KM, Castellanos A. Frequency of sudden cardiac death and profiles of risk. Am J Cardiol. 1997 Sep 11;80(5B):10F-19F. doi: 10.1016/s0002-9149(97)00477-3. PMID 9291445
- [Background] Wilson PW, D'Agostino RB, Levy D, Belanger AM, Silbershatz H, Kannel WB. Prediction of coronary heart disease using risk factor categories. Circulation. 1998 May 12;97(18):1837-47. doi: 10.1161/01.cir.97.18.1837. PMID 9603539
- [Background] Ridker PM, Rifai N, Rose L, Buring JE, Cook NR. Comparison of C-reactive protein and low-density lipoprotein cholesterol levels in the prediction of first cardiovascular events. N Engl J Med. 2002 Nov 14;347(20):1557-65. doi: 10.1056/NEJMoa021993. PMID 12432042